CLINICAL TRIAL: NCT03166033
Title: Case-control Study on Individual Risk Factors of Carpal Tunnel Syndrome
Brief Title: Case-control Study on Individual Risk Factors of CTS
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Guan Wenjie, Dr., Fudan University
Other Study IDs: 81572127
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; etiology; risk factor
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Communicable Disease Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: age between 41 and 70years. People in the case group with the symptom "numbness" and then were clinical and neural-electrophysiological diagnosed CTS. People in the control group would be exclude the symptom "numbness". The case group included clinical diagnosed carpal tunnel syndrome which was divided into 4 parts every 10 years old age. The gender of the patients of the control group was matched to the case group and divided into 4 parts by age.
  Interventions: Other: the disease
- Control Group: The present case-control study was based on the single medical center in Shanghai, China, in which more than 5000 CTS patients per year are treated. The hospital involved in the study is a university teaching hospital. Cases were recruited from the surgical wards and appropriate outpatient clinics, while the controls were recruited from the outpatient clinics. Both groups filled out a standardized questionnaire, and a standardized patient record was filled out by a hand surgeon. In addition, participants with jobs involving lifting and carrying of loads were interviewed.
  Interventions: Other: the disease

INTERVENTIONS:
Other: the disease — Observation the patients and non-patients

SUMMARY:
This study is conducted to observe the characteristics of the risk factors of CTS in Chinese population.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS), or median neuropathy at the wrist, is a medical condition in which the median nerve is compressed at the wrist, leading to paresthesia, numbness and muscle weakness in the hand. It's the most common neuro-compressive disease. With the development of the modern life, the morbidity of CTS is also raised. As a common disease, the study on etiology is very important in Carpal Tunnel Syndrome, which can improve the life quality of patients with carpal tunnel syndrome. The risk factors include individual factors such as age, gender, diabetes, Hypothyroidism, obesity, complication of systematic diseases, tobacco, injury and occupational factors.

As most of the research were based on the population in western country and the life style and the ethnicity between Chinese people and western country people is quite different, there may be some similarities and differences in epidemiology. There is seldom similar research in China so that this study was conducted to observe the characteristics of these risk factors in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* with the symptom "numbness"
* clinical and neural-electrophysiological diagnosed CTS

Exclusion Criteria:

* suffered from other diseases that could cause "numbness" diagnosed clinically

Ages: 41 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present case-control study was based on the single medical center in Shanghai, China, in which more than 5000 CTS patients per year are treated. The hospital involved in the study is a university teaching hospital. Cases were recruited from the surgical wards and appropriate outpatient clinics, while the controls were recruited from the outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 6048 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
general risk factors | 2014-2015
  Gender, age, smoking, wrist injury, diabetes mellitus, hypothyroidism and wrist working are all the risk factors of carpal tunnel syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao KM, Hu JJ, Lao J, Zhao X. Evaluation of nerve transfer options for treating total brachial plexus avulsion injury: A retrospective study of 73 participants. Neural Regen Res. 2018 Mar;13(3):470-476. doi: 10.4103/1673-5374.228730. PMID 29623932